CLINICAL TRIAL: NCT01291433
Title: Randomized Clinical Trial Evaluating Combined Pentoxifylline-tocopherol-clodronate vs Placebo in Radiation-induced Brachial Plexopathy: the PENTOCLO Trial
Brief Title: Trial of Combined Pentoxifylline-tocopherol-clodronate vs Placebo in Radiation-induced Brachial Plexopathy
Acronym: PENTOCLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P081239
Record Dates: First submitted 2011-02-02; First posted 2011-02-08 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-12

CONDITIONS: Radiation Induced Brachial Plexopathy
MeSH Terms: conditions — Radiation induced brachial plexopathy | interventions — Pentoxifylline; alpha-Tocopherol; Clodronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PENTOCLO (Experimental): Association pentoxifylline, tocopherol and clodronate
  Interventions: Drug: Pentoxifylline; Drug: Tocopherol acetate; Drug: Clodronic Acid
- Placebo (Placebo Comparator): Triple placebo
  Interventions: Drug: Pentoxifylline placebo; Drug: Tocopherol placebo; Drug: Clodronate placebo

INTERVENTIONS:
Drug: Pentoxifylline placebo — Placebo for pentoxifylline 400 mg, 1 cp twice a day (7d/7)
  Other Names: Placebo for pentoxifylline 400 mg, 1 cp twice a day (7d/7)
  Arms: Placebo
Drug: Pentoxifylline — Pentoxifylline 400 mg: 1 cp twice a day (7d/7)
  Other Names: Pentoxifylline 400 mg: 1 cp twice a day (7d/7)
  Arms: PENTOCLO
Drug: Tocopherol acetate — Tocopherol alpha-acetate, 500 mg: 1 capsule twice a day (7d/7)
  Other Names: Tocopherol alpha-acetate
  Arms: PENTOCLO
Drug: Clodronic Acid — Clodronate disodium (clodronic acid) 800 mg: 2 cp per day, 5d/7 (from monday to friday)
  Other Names: Clodronate disodium
  Arms: PENTOCLO
Drug: Tocopherol placebo — Placebo for Tocopherol alpha-acetate, 500 mg: 1 capsule twice a day (7d/7)
  Arms: Placebo
Drug: Clodronate placebo — Placebo for clodronate disodium (clodronic acid) 800 mg: 2 cp per day, 5d/7 (from monday to friday)
  Arms: Placebo

SUMMARY:
Radiation-induced brachial plexopathy (RIP) is a rare and severe delayed peripheral nerve complication of radiotherapy, that is spontaneously irreversible with no medical treatment to limit or reduce symptoms. The investigators planed in RIP a randomized double blind clinical trial, using a pentoxifylline (P)- tocopherol (E)- clodronate combination versus placebo, to assess a possible symptomatic regression by a sensory-motor neurological quantifiable and reproducible score (modified Subjective Objective Medical management Analytic, SOMA).

The investigators previously developed a successful PE treatment in symptomatic RI injuries via the antioxidant pathway, in clinical phase II and III trails and experiments obtaining a major significant radiation-induced fibrosis regression, then the PE clodronate combination (PENTOCLO), obtaining a rapid and significant healing of mandible osteoradionecrosis and significant neurological signs regression (- 35% modified SOMA score at 18 months) in 50 partial RIP.

The aim of this phase III randomized clinical trial is to show PENTOCLO efficiency and its tolerance in long survival patients irradiated before for cancer and presenting with partial RIP of upper or lower legs.

The investigators calculated to include 60 patients to show a significant clinical difference between the two groups after 18 months of treatment: PENTOCLO[Pentoxifylline 400 (2x/d) + vitamine E 500 (2x/d) + intermittent Clodronate 800 (2/d, 5d/7)] versus triple placebo, with prednisone 20 (2d/7) for all patients.

RIP is assessed before treatment and every 6 months by a standardized sensory-motor neurological (SOMA 95 modified by NCI-CTC 99) score used for main criteria at M18, and various neurological scales of assessment (Visual Analog Scale for pain / VAS for paresthesia, Neuropathic Pain Symptom Inventory [NPSI], Overall Disability Sum Score [ODSS], muscle testing, Nine hole peg test / Timed 25-Foot Walk), quality of life (SF36, Patient Global Impression of Change and Clinical Global impression of Change [PGIC/ CGIC]) and electrophysiology.

DETAILED DESCRIPTION:
The aim of this phase III randomized clinical trial is to show PENTOCLO efficiency and its tolerance in long survival patients irradiated before for cancer and presenting with partial RIP of upper or lower legs.

We calculated to include 60 patients to show a significant clinical difference between the two groups after 18 months of treatment: PENTOCLO [Pentoxifylline 400 (2x/d) + vitamine E 500 (2x/d) + intermittent Clodronate 800 (2/d, 5d/7)] versus triple placebo, with prednisone 20 (2d/7) for all patients.

RIP is assessed before treatment and every 6 months by a standardized sensory-motor neurological (SOMA 95 modified by NCI-CTC 99) score used for main criteria at M18, and various neurological scales of assessment (Visual Analog Scale [VAS] for pain / VAS for paresthesia, Neuropathic Pain Symptom Inventory [NPSI], Overall Disability Sum Score [ODSS], muscle testing, Nine hole peg test / Timed 25-Foot Walk), quality of life (SF36, Patient Global Impression of Change and Clinical Global impression of Change [PGIC/ CGIC]) and electrophysiology.

ELIGIBILITY:
Inclusion Criteria:

* Past-history of post-operative or exclusive irradiation (RT) for currently in remission cancer, in particular

  * breast cancer with breast or thoracic anterior wall RT; axilla-subclavicular lymph nodes RT; sometimes lung or head/neck cancer
  * Lymphoma (Hodgkin or non Hodgkin) with axilla-subclavicular RT (upper limb) or lumbar-aortic (lower limbs) or testis tumor
* Delay RT-RIP more than 6 months, but partial RIP
* Neurological injury in irradiated volume confirmed by EMG
* Patient living within distance compatible with day-hospitalization
* Use of effective contraception for fertile women
* Signed written informed consent (in case of motor paralysis informed consent is signed by a witness)

Exclusion Criteria:

* Localized or metastatic cancer recurrence (axillar MRI or PET scan)
* Complete plexus injury with total motor paralysis of upper/ lower limb for more than 2 years
* Associated neurological disease that may interferer with the assessment of endpoints
* Hemorrhage, disease with hemorrhagic risk, unbalanced diabetes
* Known hypersensitivity to Pentoxifylline, one of the excipients or biphosphonates
* Renal failure, liver failure or decompensated heart failure
* Taking another biphosphonate
* Evolving virosis (hepatitis, herpes, zona) or live vaccine (influenza)
* Uncontrolled psychotic condition
* Informed consent not obtained
* Fertile women who do not want or cannot use effective contraception during the administration of study drugs
* Women pregnant or nursing

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2011-03; Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Sensory-motor neurological clinical assessment | 18 months
  Sensory-motor neurological clinical assessment of RIP patients as measured with SOMA scale (Subjective Objective Medical management Analytic involving tools) modified by NCI-CTC99 scale

SECONDARY OUTCOMES:
Pain VAS | 6, 12, 18 months
  Visual analog scale for pain
NPSI scale | 6, 12, 18 months
  NPSI (Neuropathic Pain Symptom Inventory) pain scale to assess neuropathic pain by a self-questionnaire [Reference: Bouhassira et al. Development and validation of the neuropathic pain symptom inventory. Pain 2004;108(3):248-57]
Paresthesia VAS | 6, 12, 18 months
  Visual analog scale for paresthesia
Frequence of paresthesia | 6, 12, 18 months
  Evaluated on a 4-item scale:
  * Never
  * Occasional (several times each week or month)
  * Intermittent (several times a day)
  * Permanent (all day long and night)
ODSS | 6, 12, 18 months
  Overall disability sum score: Checklist for upper limb (5 items) and lower limb (7 items)
Muscle testing | 6, 12, 18 months
  Semi-quantitative manual muscle strength assessment on a 0 to 5 scale, separately for each muscle.
Neurological examination | 6, 12, 18 months
  Evaluation of sensitivity, motricity and reflex
Motor assessment of complex movements | 6, 12, 18 months
  Evaluated by two separate tests according to upper vs lower limb involvement:
  * Nine Hole Peg test for brachial injury
  * Timed 25-Foot Walk for lower limb symptoms
Quality of life | 6, 12, 18 months
  Global quality of life as evaluated by SF36 questionnaire
Global clinical impression | 6, 12, 18 months
  Patient global impression of change (PGIC) and clinical global impression of change (CGIC)
Electromyography | 6, 12, 18 months
  Electromyography of upper / lower limbs
Clinical symptoms evaluation | 6, 12, 18 months
  Clinical evaluation looking for upper digestive disorders (nausea, vomiting, epigastralgia), lower digestive disorders (diarrhea), vascular disorders (cephalalgia, vertigo, flush, deep asthenia), bleeding (hematoma)
Biological evaluation | 6, 12, 18 months
  evaluation of biological parameters: blood cell count, platelets, sedimentation velocity, C-reactive protein, prothrombin time, TCK, calcemia, protidemia, LDH, creatininemia, phosphokinase creatine (CPK)
Cardiovascular evaluation | 6, 12, 18 months
  As evaluated by:
  * Heart rate
  * Blood pressure lying and standing after 5 minutes orthostatism
  * Electrocardiogramm

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Delanian, MD, PhD, Principal Investigator — Oncologie-Radiothérapie, Hôpital Saint Louis , Paris, France
Locations (2):
- France (2):
  - Groupe Hospitalier Pitié-Salpêtrière, Paris
  - Hôpital Saint-Louis, Paris

REFERENCES:
- [Derived] Pradat PF, Maisonobe T, Psimaras D, Lenglet T, Porcher R, Lefaix JL, Delanian S. [Radiation-induced neuropathies: collateral damage of improved cancer prognosis]. Rev Neurol (Paris). 2012 Dec;168(12):939-50. doi: 10.1016/j.neurol.2011.11.013. Epub 2012 Jun 27. French. PMID 22742890